CLINICAL TRIAL: NCT01491555
Title: Electrical Impedance Myography and Ultrasound as Biomarkers of Duchenne Muscular Dystrophy
Acronym: QED
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Basil Darras, Basil Darras, M.D., Boston Children's Hospital
Other Study IDs: IRB-P00001218
Record Dates: First submitted 2011-12-05; First posted 2011-12-14 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy; DMD; controls; EIM; QUS
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- DMD patients: 35 boys ages 2 through 30 with DMD
- Control Group: 35 healthy boys ages 2 through 30

SUMMARY:
Researchers at Children's Hospital Boston Neurology Department invite children to participate in a new research study. Researchers are looking for boys ages 2 - 30 with Duchenne Muscular Dystrophy (DMD) and healthy boys ages 2 - 30 (without any nerve or muscle concerns) to serve as controls. The study is evaluating a new technique that will test nerve and muscle function. The testing is all pain free.

Children participating in the study will come in for 10 visits over two years. Visits will take place every month at first, then less often for the remaining visits. The tests for the study itself take approximately 2hours. If participants are interested or would like to learn more about the study, please call Lavanya Madabusi at 617-919-3554 or Lavanya.Madabusi@childrens.harvard.edu. All inquiries will be kept strictly confidential.

DETAILED DESCRIPTION:
Characterized by progressive disability leading to death, Duchenne muscular dystrophy (DMD) remains one of the most common and devastating neuromuscular disorders of childhood. Although a variety of promising new treatment strategies are in development, outcome measures for clinical trials remain limited for the most part to a set of functional measures, such as the six-minute walk test. While clearly useful, such measures are impacted by unrelated factors, such as mood and effort, and have limited repeatability. To address this and other limitations, magnetic resonance imaging (MRI) is now being investigated as a surrogate measure. However, more easily applied, cost-effective, office-based surrogate measures that provide high repeatability and sensitivity while still correlating strongly to disease status would find wider use in Phase II and possibly in Phase III clinical trials in DMD. Quantitative ultrasound (QUS) and electrical impedance myography (EIM) are two techniques that could serve in this role. In QUS, muscle pathology (fibrosis and fatty infiltration) in DMD results in an increase in energy reflected back (backscatter) to the ultrasound. The amount of backscatter can be measured directly by analyzing the raw frequency-based acoustic data or indirectly by controlled processing of the gray-scale image. EIM, in contrast, relies upon the application of localized electrical current and measurement of the resulting surface voltages, but is similarly impacted by the fibrotic changes that develop as muscle disease progresses. Here, the investigators propose to evaluate and compare both methodologies simultaneously in a group of DMD patients and normal subjects in order to assess their ability to identify clinically meaningful alterations in muscle health over short intervals of time. As a final exploratory analysis, the investigators will also study the possibility of combining the two modalities. The results of this work will have broad application as they could be applied to a variety of neuromuscular conditions, including other muscular dystrophies. Thus, the hypothesis of this proposal is that both QUS and EIM can serve as convenient, non-invasive, clinically meaningful surrogate markers of disease progression in DMD that surpass the functional measures currently in use.

ELIGIBILITY:
Inclusion criteria (DMD):

1. Genetically or histologically established diagnosis of DMD
2. Male, age 2 - 30

Inclusion criteria (Control):

1. Male, age 2 - 30

Exclusion criteria (DMD):

1. Presence of implanted pacemaker or other electrical device
2. Presence of a superimposed neuromuscular or other medical condition that substantially impacts the individual's health

Exclusion criteria (control):

1. Presence or past history of a neuromuscular disorder or other disease that substantially impacts health
2. Presence of implanted pacemaker or other electrical device.

Ages: 2 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This study will involve boys with DMD and healthy male controls.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2012-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
The rate of decline of DMD patients versus normal subjects as assessed by EIM and quantitative ultrasound | up to 45 months
  With the successful completion of this aim, the investigators will establish that alterations in both EIM and QUS provide meaningful surrogate measures of disease progression in DMD.

SECONDARY OUTCOMES:
The rate of decline of DMD patients versus normal subjects as assessed by handheld dynamometry, 6-minute walk, and other functional tests. | up to 45 months
  With the successful completion of this aim, the investigators will establish that alterations in functional assessments may provide additional meaningful surrogate measures of disease progression in DMD.

CONTACTS AND LOCATIONS:
Overall Officials: Basil Darras, MD, Principal Investigator — Boston Children's Hospital; Seward Rutkove, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided